CLINICAL TRIAL: NCT03104465
Title: Adaptation of Mindfulness Training to Treat Chronic Pain in the Military
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R34AT008423-01 (NIH)
Record Dates: First submitted 2017-04-03; First posted 2017-04-07 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Mindfulness; Behavioral Health; Quality of Life
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness training (Experimental): 6 90-minute sessions interactive, web-based mindfulness training complemented with mobile application
  Interventions: Behavioral: Mindfulness Training

INTERVENTIONS:
Behavioral: Mindfulness Training — interactive. web-based mindfulness training complemented with mobile application

SUMMARY:
The overall aim of this study is to test the acceptability and feasibility of an interactive, web-based mindfulness training with active duty soldiers being treated for chronic pain.

DETAILED DESCRIPTION:
The overall aim of study is to test the acceptability and feasibility of an interactive, web-based mindfulness training with active duty soldiers being treated for chronic pain. We will adapt the evidence-based Mindfulness-based Stress Reduction (MBSR) training for use with this population. The adapted training will be enhanced by mobile applications (apps) for skills practice, using an existing apps platform.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who have experienced chronic pain for at least 6 months

Exclusion Criteria:

* Do not have any of the following conditions: substance abuse or dependence, psychosis, suicidal ideation in the last 2 months, high levels of trauma symptoms,
* plans to have a permanent change of station or deploy in the coming 6 months, or
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2018-06-11 (Actual)

PRIMARY OUTCOMES:
Chronic Pain - Pain Intensity | Baseline
  Assess pain intensity using the Patient Reported Outcomes Measurement Information System (PROMIS) Short Form (SF) v.1.0 - Pain Intensity 3a
Chronic Pain - Pain Intensity | 6 - 8 weeks post-treatment
  Assess pain intensity using the Patient Reported Outcomes Measurement Information System (PROMIS) Short Form (SF) v.1.0 - Pain Intensity 3a
Chronic Pain - Pain Interference | Baseline
  Assess pain intensity using the Patient Reported Outcomes Measurement Information System (PROMIS) Short Form (SF) v.1.0 - Pain Interference 8a
Chronic Pain - Pain Interference | 6 - 8 weeks post-treatment
  Assess pain intensity using the Patient Reported Outcomes Measurement Information System (PROMIS) Short Form (SF) v.1.0 - Pain Interference 8a
Chronic Pain | Baseline
  Assess intensity of sensory and affective pain using Short-Form McGill Pain Questionnaire
Chronic Pain | 6 - 8 weeks post-treatment
  Assess intensity of sensory and affective pain using Short-Form McGill Pain Questionnaire

SECONDARY OUTCOMES:
Co-Occurring Conditions - Depression | Baseline
  Assess depression using Patient Reported Outcomes Measurement Information System (PROMIS) Short Form (SF) v.1.0 - Emotional Distress - Depression 8a
Co-Occurring Conditions - Depression | 6 - 8 weeks post-treatment
  Assess depression using Patient Reported Outcomes Measurement Information System (PROMIS) Short Form (SF) v.1.0 - Emotional Distress - Depression 8a
Co-Occurring Conditions - Anxiety | Baseline
  Assess anxiety using Patient Reported Outcomes Measurement Information System (PROMIS) Short Form (SF) v1.0 - Emotional Distress- Anxiety 6a
Co-Occurring Conditions - Anxiety | 6 - 8 weeks post-treatment
  Assess anxiety using Patient Reported Outcomes Measurement Information System (PROMIS) Short Form (SF) v1.0 - Emotional Distress- Anxiety 6a
Co-Occurring Conditions - Alcohol Use | Baseline
  Assess hazardous and harmful alcohol use and dependence using the Alcohol Use Disorders Identification Test (AUDIT)
Co-Occurring Conditions - Alcohol Use | 6 - 8 weeks post-treatment
  Assess hazardous and harmful alcohol use and dependence using the Alcohol Use Disorders Identification Test (AUDIT)
Co-Occurring Conditions - Post Traumatic Stress Disorder | Baseline
  Assess trauma symptoms in response to stressful experiences using the Post Traumatic Stress Disorder (PTSD) Checklist - Civilian version (PCL-C)
Co-Occurring Conditions - Post Traumatic Stress Disorder | 6 - 8 weeks post-treatment
  Assess trauma symptoms in response to stressful experiences using the Post Traumatic Stress Disorder (PTSD) Checklist - Civilian version (PCL-C)
Co-Occurring Conditions - Prescription drug misuse | Baseline
  Assess use of drugs not prescribed, or use of more than recommended dose, to feel good/get high/buzzed
Co-Occurring Conditions - Prescription drug misuse | 6 - 8 weeks post-treatment
  Assess use of drugs not prescribed, or use of more than recommended dose, to feel good/get high/buzzed
Quality of Life - Physical Functioning | Baseline
  Assess physical functioning using Patient Reported Outcomes Measurement Information System (PROMIS) Short Form (SF) v.1.0 - Physical Function 12a
Quality of Life - Physical Functioning | 6 - 8 weeks post-treatment
  Assess physical functioning using Patient Reported Outcomes Measurement Information System (PROMIS) Short Form (SF) v.1.0 - Physical Function 12a
Quality of Life - Sleep disturbance | Baseline
  Assess sleep quality, depth and restoration using Patient Reported Outcomes Measurement Information System (PROMIS) Short Form (SF) v.1.0 - Sleep Disturbance 8a
Quality of Life - Sleep disturbance | 6 - 8 weeks post-treatment
  Assess sleep quality, depth and restoration using Patient Reported Outcomes Measurement Information System (PROMIS) Short Form (SF) v.1.0 - Sleep Disturbance 8a
Quality of Life - Fatigue | Baseline
  Assess fatigue using Patient Reported Outcomes Measurement Information System (PROMIS) Short Form (SF) v.1.0 - Fatigue 8a
Quality of Life - Fatigue | 6 - 8 weeks post-treatment
  Assess fatigue using Patient Reported Outcomes Measurement Information System (PROMIS) Short Form (SF) v.1.0 - Fatigue 8a
Quality of Life - Role satisfaction | Baseline
  Assess social satisfaction using Patient Reported Outcomes Measurement Information System (PROMIS) Short Form (SF) v.1.0 - Ability to Participate in Social Roles & Activities 8a
Quality of Life - Role satisfaction | 6 - 8 weeks post-treatment
  Assess social satisfaction using Patient Reported Outcomes Measurement Information System (PROMIS) Short Form (SF) v.1.0 - Ability to Participate in Social Roles & Activities 8a
Self-Regulation - Pain Catastrophizing Scale | Baseline
  Assess experience of pain through sub-scales of rumination, magnification and helplessness
Self-Regulation - Pain Catastrophizing Scale | 6 - 8 weeks post-treatment
  Assess experience of pain through sub-scales of rumination, magnification and helplessness
Self-Regulation - Chronic Pain Acceptance Scale | Baseline
  Assess behavioral aspects of chronic pain acceptance
Self-Regulation - Chronic Pain Acceptance Scale | 6 - 8 weeks post-treatment
  Assess behavioral aspects of chronic pain acceptance
Self-Regulation - Emotional Behavioral Dysregulation | Baseline
  Assess emotional behavioral dysregulation using Patient Reported Outcomes Measurement Information System (PROMIS) Short Form (SF) v.1.0 - Emotional and Behavioral Dyscontrol
Self-Regulation - Emotional Behavioral Dysregulation | 6 - 8 weeks post-treatment
  Assess emotional behavioral dysregulation using Patient Reported Outcomes Measurement Information System (PROMIS) Short Form (SF) v.1.0 - Emotional and Behavioral Dyscontrol
Mindfulness | Baseline
  Assess mindfulness using the Five Factor Mindfulness Questionnaire (FFMQ)
Mindfulness | 6 - 8 weeks post-treatment
  Assess mindfulness using the Five Factor Mindfulness Questionnaire (FFMQ)

CONTACTS AND LOCATIONS:
Overall Officials: Shari Miller, PhD, Principal Investigator — RTI International
Locations (1):
- Womack Army Medical Center at Ft. Bragg, Fort Bragg, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No